CLINICAL TRIAL: NCT02603055
Title: A Phase Ib Single Center, Randomized, Blinding, Parallel-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of a Recombinant Hepatitis E Vaccine in Healthy Adults Aged 16 to 65 Years Old in China
Brief Title: A Clinical Trial to Evaluate a Recombinant Hepatitis E Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Changchun Institute of Biological Products Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JSVCT025
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis E
Keywords: Safety; immunogenicity; Hepatitis E
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30μg/0.5ml Hepatitis E vaccine (Experimental): three doses, 30μg/0.5ml per dose
  Interventions: Biological: 30μg/0.5ml Hepatitis E vaccine
- 30μg/0.5ml Recombinant Hepatitis E vaccine (Active Comparator): 30μg/0.5ml Hepatitis E vaccine developed by Xiamen innovax biotech Co., Ltd. three doses, 30μg/0.5ml per dose
  Interventions: Biological: 30μg/0.5ml Recombinant Hepatitis E vaccine

INTERVENTIONS:
Biological: 30μg/0.5ml Hepatitis E vaccine — three doses, 30μg/0.5ml per dose
  Arms: 30μg/0.5ml Hepatitis E vaccine
Biological: 30μg/0.5ml Recombinant Hepatitis E vaccine — 30μg/0.5ml Hepatitis E vaccine developed by Xiamen innovax biotech Co.,Ltd.,three doses, 30μg/0.5ml per dose
  Arms: 30μg/0.5ml Recombinant Hepatitis E vaccine

SUMMARY:
Hepatitis E is characteristic by sporadic and local epidemic around the world, and mainly infects adults aged 15 to 40 years old, resulting in the infection rate ranged from 1% to 15%. The investigational hepatitis E vaccine is a recombinant aluminium-adjuvant hepatitis E vaccine.

This is a single center, randomized, blinding, parallel-controlled phase Ib clinical trial. This study will determine the safety and immunogenicity of the investigational recombinant hepatitis E vaccine in healthy adults between 16 and 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 and 65 years with normal intelligence.
* Negative in antibody against hepatitis E test.
* No plan to go out for a long time within 9 months.
* Able to understand the content of informed consent and willing to sign the informed consent
* General good health as established by medical history and physical examination.
* Able and willing to complete all the secluded study process during the whole study follow-up period.
* No history of hepatitis B, hepatitis C and hepatitis E(Patients diagnosed as hepatitis B, hepatitis C and hepatitis E by town or above)
* Axillary temperature ≤37.0°C on the day of enrollment

Exclusion Criteria:

* Woman who is pregnant, breast-feeding or planning to be pregnant during the study period
* Allergic history of any vaccination or drugs, or allergic to any ingredient of the Hepatitis E vaccine
* History of serious adverse reactions after vaccination, such as allergies, urticaria, breathing difficulties, angioneurotic oedema or abdominal pain
* Autoimmune disease or immunodeficiency
* Asthma that was unstable and need emergency treatment, hospitalization, oral or intravenous corticosteroid within two years
* Type I or II diabetes, not including gestational diabetes
* History of thyroidectomy, or need treatment for thyroid disease in the past 12 months
* History of serious angioneurotic edema in the past 3 years, or need treatment for it in the past 2 years
* Severe hypertension, with the blood pressure still more than 150/100 mmHg after drug maintenance treatment
* Abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or coagulation disorders diagnosed by the doctor.
* Patients who are active or not have a definite cure of malignant tumors, or who may recur in the study period.
* Epilepsy, not including alcohol epilepsy in the first 3 years abstinence or simple epilepsy without the need of treatment in the past 3 years
* Asplenia or functional asplenia, or asplenia and splenectomy under any circumstances
* Guillain Barre Syndrome
* Prior administration of immunodepressant, cytotoxic or corticosteroids (not including corticosteroid therapy for allergic rhinitis and acute non concurrent dermatitis )treatment in last 6 months
* Prior administration of immune globulin in last 3 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine in last 1 month
* Prior administration of subunit or inactivated vaccine in last 14 days, such as pneumococcal Vaccine
* Current anti-tuberculosis prophylaxis or therapy
* Fever (axillary temperature 38.0℃) in 3 days before vaccination or any acute disease, systemic application of antibiotics or antiviral therapy in the past five days
* Unable to comply with the study requirements due to the psychological situation, a past or present history of mental disease, two-stage affective psychosis which were not well controlled in the past two years; mental disease need medical treatment, and have suicidal tendency over the past five years
* Any condition that in the opinion of the investigators may interfere with the evaluation of study objectives

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse reactions after vaccination | within 7 days after each vaccination
  Occurrence of adverse reactions within 7 days after each vaccination with the Recombinant Hepatitis E vaccine.
The geometric mean concentration of antibody against Hepatitis E responses to the Hepatitis E vaccine | 7 months after the first vaccination
  Antibody against Hepatitis E responses to the Hepatitis E vaccine at 7 months after the first vaccination

SECONDARY OUTCOMES:
Occurrence of adverse events after each vaccination | within 28 days after each vaccination
  Occurrence of adverse events within 28 days after each vaccination with the Hepatitis E vaccine.
Occurrence of serious adverse events after the vaccination. | within 12 months after the first vaccination
  Occurrence of serious adverse events within 12 months after the first vaccination with the Hepatitis E vaccine.
The positive rates of antibody against Hepatitis E responses to the Hepatitis E vaccine. | 7 months after the first vaccination
  The positive rates of antibody against Hepatitis E responses to the Hepatitis E vaccine at 7 months after the first vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China